CLINICAL TRIAL: NCT04375475
Title: Evaluation of the Effect of Changyou Probiotic Flavored Yogurt on Intestinal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bright Dairy & Food Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19-SM-02-GM-001
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Intestinal Health

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bright Changyou probiotic flavored yogurt (Experimental): Bright Changyou probiotic flavored yogurt contains 5.0×10^8cfu/g of probiotics including Lactobacillus bulgaricus, Streptococcus thermophilus, Bifidobacterium lactis, Lactobacillus acidophilus, Lactobacillus plantarum ST-Ⅲ (7mg/kg), and 1.5% of inulin
  Interventions: Dietary Supplement: Bright Changyou probiotic flavored yogurt
- Bright Changyou lactobacillus flavored yogurt (Active Comparator): Bright Changyou flavored yogurt contains probiotics including Lactobacillus bulgaricus, Streptococcus thermophilus, Bifidobacterium lactis, Lactobacillus acidophilus, and Lactobacillus plantarum ST-Ⅲ (7mg/kg)
  Interventions: Dietary Supplement: Bright Changyou lactobacillus flavored yogurt
- Bright flavored yogurt (Active Comparator): Bright flavored yogurt contains Lactobacillus bulgaricus, Streptococcus thermophilus, Lactobacillus acidophilus, Bifidobacterium lactis, and Lactobacillus casei LC2W (0.1 mg/kg)
  Interventions: Dietary Supplement: Bright flavored yogurt

INTERVENTIONS:
Dietary Supplement: Bright Changyou probiotic flavored yogurt — Oral consumption of Bright Changyou probiotic flavored yogurt 100 g at a time and twice per day for 28 days. The experimental product has similar package and taste as the comparators.
  Arms: Bright Changyou probiotic flavored yogurt
Dietary Supplement: Bright Changyou lactobacillus flavored yogurt — Oral consumption of Bright Changyou lactobacillus flavored yogurt 100 g at a time and twice per day for 28 days.
  Arms: Bright Changyou lactobacillus flavored yogurt
Dietary Supplement: Bright flavored yogurt — Oral consumption of Bright flavored yogurt 100 g at a time and twice per day for 28 days.
  Arms: Bright flavored yogurt

SUMMARY:
This was a randomized, double-blind, single-center, placebo-controlled, three-arm study.

The objectives of this study were to evaluate the effect of the Bright Changyou Probiotic Flavored Yogurt on:

Improving gastrointestinal health; Relieving symptoms of functional constipation or functional diarrhea; Improving gut immunity; Adjusting microbiological flora in gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 25-45 years old;
* Functional constipation or diarrhea diagnosed by Rome III criteria;
* Agree not to take any dietary supplements or dairy products other than the study products during the study period;
* Agree not to take any supplements or dairy products containing prebiotics/probiotics other than the study products during the study period;
* Agree not to participant in other interventional studies during the study period;
* Fully understand the property, purpose, benefits and potential risk and side effect from the study;
* Agree to follow all study requirements and procedures;
* Signed informed consent.

Exclusion Criteria:

* Currently receiving treatment for gastrointestinal symptoms;
* Lactose intolerance;
* Having diseases or conditions that may affect intestinal function, such as history of gastrointestinal resection, colon or rectal cancer, inflammatory bowel disease, diabetes, hyperthyroidism or hypothyroidism, Hirschsprung's disease, scleroderma, or Anorexia nervosa;
* Currently under diet control or in use of medicine or supplements for weight control or that might affect appetite;
* Have had laxatives or other substance that will enhance digestion within two weeks before the study begins;
* Have had dairy products or other food containing probiotics within 10 days before the study begins;
* Currently having diarrhea;
* Currently pregnant or breast-feeding, or plan to be pregnant during the study period;
* Not be able to follow study procedures according to investigators evaluation.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 198 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal health score | Day 0, 28
  Change of the total gastrointestinal health score at day 28 from baseline. The total score is the sum of the 4 aspects of gastrointestinal health (each with score range from 0 to 3):
  Weekly stool frequency (>=6; 4-6; 1-3; 0); Ratio of the number of unopened defecation to the total number of defecation (1; 1/4; 1/3; >=1/2); Duration of defecation (<5 minutes; 5-15 minutes; 16-30 minutes; >=30 minutes); Defecation condition (normal perception; straining/uncomfortableness at stool; obvious straining/uncomfortableness or difficulty at defecation with little feces amount; frequent abdominal or anus pain that affect defecation).

SECONDARY OUTCOMES:
Defecation satisfaction score | Day 0, 3, 7, 14, 21, 28
  Total score of the satisfaction on 4 aspects of defecation habit (each with score range from 0 to 3):
  Stool frequency, defecation duration, stool characteristics, and defecation habit (very satisfied; satisfied; neither satisfied nor dissatisfied; dissatisfied)
Bristol score of stool characteristics | Day 0, 3, 7, 14, 21, 28
  1. Separate hard lumps, like nuts;
  2. Sausage-shaped but lumpy;
  3. Like a sausage but with cracks on the surface;
  4. Like a sausage or snake, smooth and soft;
  5. Soft blobs with clear-cut edges;
  6. Fluffy pieces with ragged edges, a mushy stool;
  7. Watery, no solid pieces, entirely liquid.
Bristol score of stool color | Day 0, 3, 7, 14, 21, 28
  Score from 1 to 7 for stool color from light to dark
Symptom score of digestive system | Day 0, 3, 7, 14, 21, 28
  Total score of the 9 aspects of digestive symptoms (each with score range from 0 to 3 indication no symptom, light symptom, moderate symptom and severe symptom):
  Bloating, abdominal pain, gastric distention, heavy stomach, loss of appetite, belching, intestinal colic, and abdominal colic.
Fecal bacterium | Day 0, 14
  Quantitative measurements of clostridium perfringens bacteria, lactobacillus, bifidobacterium and Escherichia coli.
Fecal short chain fatty acids | Day 0, 14
  Percentage of acetic acid, propionic acid and butyric acid
Fecal secretory immunoglobulin A (sIgA) | Day 0, 14
  Fecal concentration of sIgA

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaoton University Affiliated Xinhua Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No